CLINICAL TRIAL: NCT04579172
Title: Cervico-Isthmic Compression Suture Versus Anterior Wall Uterine Resection in Cases of Morbidly Adherent Anterior Situated Placenta
Brief Title: Conservative Management of Morbidly Adherent Anterior Situated Placenta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Taman, lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS.20.09.1246
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: - Randomized controlled trial (RCT) of pregnant women recruited from Department of Obstetrics and Gynecology Mansoura University Hospitals for elective termination of pregnancy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Circular isthmic-cervical sutures
  Interventions: Procedure: Cervico- isthmic compression suture
- Group B (Experimental): Resection of the infiltrated part of anterior uterine wall
  Interventions: Procedure: Anterior wall uterine resection:

INTERVENTIONS:
Procedure: Cervico- isthmic compression suture — Circular isthmic-cervical sutures will be applied . To avoid ureter and bladder injury, the bladder will be reflected downward. A silastic drain will be inserted into internal and through the external os , so as to drain the uterine cavity and to keep the cervical canal open. Firstly, at the left side of the uterus, a Vicryl number two (No..2) stitch will be inserted very close to the cervix from the anterior to the posterior side of the broad ligament.
  Arms: Group A
Procedure: Anterior wall uterine resection: — After fetal delivery, two corners of the uterine incision and the superior and inferior lips will be clamped immediately by four Mayo clamps. Blunt dissection downward to the bladder-uterus peritoneal reflection will perform, to the partial anterior wall of the uterine myometrium where the placenta was deeply adherent (a myometrium defect, with only the serous layer of the uterus) will be respected, together with the placenta. It is important to ensure that sufficient myometrium above the peritoneal reflection will be available for an optimum closure. Then, as much remaining placenta as possible will be removed piecemeal from the edge of the uterine incision. Clamps and multiple hemostatic sutures will be applied rapidly
  Arms: Group B

SUMMARY:
Placenta accreta is defined as abnormal trophoblast invasion of part or the entire placenta into the myometrium of the uterine wall. Placenta accreta spectrum (PAS), formerly known as morbidly adherent placenta, refers to the range of pathologic adherence of the placenta, including placenta increta, percreta, and accreta.

An important risk factor of placenta accreta is placenta previa in the presence of a uterine scar. Placenta previa is an independent risk factor for placenta accreta.Additional reported risk factors for placenta accreta include increased maternal age and multiparity, other prior uterine surgery, prior uterine curettage,uterine irradiation, Asherman syndrome, uterine leiomyomata, uterine anomalies, hypertensive disorders of pregnancy and smoking. (1,2) Maternal morbidity and mortality can occur because of severe and sometimes life-threatening hemorrhage, which often requires blood transfusion also and rates of maternal death are increased for women with PAS. Additionally, patients with PAS are more likely to require hysterectomy at the time of delivery or during the postpartum period and have longer hospital stays states.(3) According to FIGO Classification of PAS Disorders 2019 There are three grades. Grade 1: abnormally adherent placenta (placenta adherent or accreta) - attached directly to the surface of the middle layer of the uterine wall (myometrium) without invading it, Grade 2: abnormally invasive placenta (increta) - invasion into the myometrium and Grade 3: abnormally invasive placenta (percreta) invasion may reach surrounding pelvic tissues, vessels and organs.(4) Nowadays, fertility sparing and conservative methods can be applied. These methods include placenta left in situ, cervical inversion technique , triple-P procedure, cervico-isthmic compression suture and anterior wall uterine resection

DETAILED DESCRIPTION:
Study Design & Area:

Randomized controlled trial (RCT) of pregnant women recruited from Department of Obstetrics and Gynecology Mansoura University Hospitals during September 2020 until September 2021 and may be extended if needed.

The study groups will undergo:

Informed consent

History:

Personal: (age, duration of marriage, special habits). Menstrual history Obstetric: (parity, mode of delivery, fetal outcome). Present history of any medical or obstetric problems. Past medical and surgical history. Clinical examination : General and obstetric examination

Calculation of Gestational Age :

Gestational age will be calculated by adding 280 days (40weeks) to the first day of the last menstrual period or by ultrasound.

Investigation:

Lab investigation:- Complete blood count , Bleeding profile, international normalization ratio, liver function tests, kidney function tests

Ultrasound:

Ultrasound Finding:- i. Establish the presence of a living fetus. ii. Estimate the age of the pregnancy. iii. Diagnose congenital abnormalities of the fetus. iv. Evaluate the position of the fetus. v. Determine the amount of amniotic fluid around the baby. vi. Assess fetal growth. vii. Assess fetal well-being. viii. Evaluate the position of the placenta.

- When the antepartum diagnosis of placenta accreta is made, it is usually based on ultrasound findings in the second or third trimester. Sonographic findings that may be suggestive of placenta accreta include:

1. Loss of normal hypoechoic retroplacental zone.
2. Multiple vascular lacunae (irregular vascular spaces) within placenta, giving "Swiss cheese" appearance.
3. Blood vessels or placental tissue bridging uterine-placental margin, myometrial-bladder interface.
4. Retroplacental myometrial thickness of <1 mm. 3 - Color Doppler criteria:

   * Diffuse or focal lacunar flow pattern.
   * Sonolucent vascular lakes with turbulent flow typified by high-velocity (peak systolic velocity>15 cm/s) and low-resistance waveform.
   * Markedly dilated vessels over the peripheral subplacental region (6)

Surgical Procedure:

Preparation of the patient before surgery:

* Patient will shave their pubic hair , take a shower with an antiseptic soap, antibiotic prophylaxis and urinary catheter insertion .
* Caesarean section steps :

After spinal anesthesia and skin sterilization Abdominal Incision: Pfannenstiel incision then cut the subcutaneous fat and rectus sheath and blunt entry into the peritoneal cavity .

ELIGIBILITY:
Inclusion Criteria:

* 1- Patient with FIGO classification of PAS disorders Grade 1 & Grade 2 which diagnosed by :

  1. Loss of normal hypoechoic retroplacental zone.
  2. Multiple vascular lacunae (irregular vascular spaces) within placenta, giving "Swiss cheese" appearance.
  3. Retroplacental myometrial thickness of less 1 mm. 2- Patient welling to preserve fertility.

Exclusion Criteria:

* 1- Patient with FIGO classification of PAS disorders Grade 3 (interruption of the hyperechoic border between the uterine serosa and bladder by US).

  2- Age : >40 years old. 3- Patient has medical disorders: cardiac disease, uncontrolled DM, chronic renal disease, chronic liver disease.

  4- Patient who refuse to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females diagnosed to have placenta Previa or morbidly adherent placenta
Enrollment: 40 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
estimated blood loss | from the start of uterine incision till closure of uterine wall
  1. The amount of blood drawn into the storage jar during surgery (suction apparatus).
  2. The weight of blood-soaked gauze pads, gauzes, and surgical dressings minus their preoperative weight, and corresponding conversion according to the proportion of 1.05 g in weight to 1 ml in volume.

SECONDARY OUTCOMES:
hemoglobin deficit | from the induction of anesthesia till 2 hours after the end of surgery
  Compare hemoglobin and hematocrit values before and after operation.
complication rate | from the start of induction of anesthesia till 24 hours after the end of surgery
  1. Injury to local organs (e.g., bowel, bladder, uterus and neurovascular structures in the retroperitoneum and lateral pelvic sidewalls from placental implantation and its removal).
  2. Postpartum hemorrhage, Internal hemorrhage.
  3. Amniotic fluid embolism.
  4. Massive blood transfusion: acidosis, hypothermia, coagulopathy, electrolyte abnormalities and infection.
  5. Postoperative thromboembolism, infection, multisystem organ failure, and maternal death
  6. Hysterectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauniaux E, Ayres-de-Campos D, Langhoff-Roos J, Fox KA, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO classification for the clinical diagnosis of placenta accreta spectrum disorders. Int J Gynaecol Obstet. 2019 Jul;146(1):20-24. doi: 10.1002/ijgo.12761. PMID 31173360
- [Background] Jauniaux E, Kingdom JC, Silver RM. A comparison of recent guidelines in the diagnosis and management of placenta accreta spectrum disorders. Best Pract Res Clin Obstet Gynaecol. 2021 Apr;72:102-116. doi: 10.1016/j.bpobgyn.2020.06.007. Epub 2020 Jun 27. PMID 32698993
- [Background] Zhao X, Tao Y, Du Y, Zhao L, Liu C, Zhou Y, Wei P. The application of uterine wall local resection and reconstruction to preserve the uterus for the management of morbidly adherent placenta: Case series. Taiwan J Obstet Gynecol. 2018 Apr;57(2):276-282. doi: 10.1016/j.tjog.2018.02.017. PMID 29673673